CLINICAL TRIAL: NCT04672083
Title: A Phase Ia Clinical Study of HIV Entry Inhibitor CPT31: Single Ascending Dose Study of Safety, Tolerability, Immunogenicity, and Pharmacokinetics in Healthy Adults
Brief Title: A Clinical Study of the HIV Drug CPT31 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Navigen, Inc. (Industry)
Collaborators: Covance (Industry); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPT31-001; 2U44AI095172-08 (NIH)
Record Dates: First submitted 2020-12-08; First posted 2020-12-17 (Actual); Results first posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-01

CONDITIONS: HIV Infections
Keywords: D-peptide HIV entry inhibitor
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): 6 subjects receiving a single subcutaneous injection of CPT31 (0.01 mg/kg) and 2 subjects receiving matching placebo SC injection
  Interventions: Drug: CPT31; Drug: Placebo
- Cohort 2 (Experimental): 6 subjects receiving a single subcutaneous injection of CPT31 (0.04 mg/kg) and 2 subjects receiving matching placebo SC injection
  Interventions: Drug: CPT31; Drug: Placebo
- Cohort 3 (Experimental): 6 subjects receiving a single subcutaneous injection of CPT31 (0.12 mg/kg) and 2 subjects receiving matching placebo SC injection
  Interventions: Drug: CPT31; Drug: Placebo
- Cohort 4 (Experimental): 6 subjects receiving a single subcutaneous injection of CPT31 (0.24 mg/kg) and 2 subjects receiving matching placebo SC injection
  Interventions: Drug: CPT31; Drug: Placebo

INTERVENTIONS:
Drug: CPT31 — CPT31 (cholesterol-PIE12-2-trimer) is a novel D-peptide HIV entry inhibitor that binds with high affinity to a conserved hydrophobic pocket within the gp41 trimer
  Other Names: cholesterol-PIE12-2-trimer; cholesterol-PIE12-trimer
Drug: Placebo — matching placebo

SUMMARY:
This first-in-human study will evaluate the safety, tolerability, immunogenicity, and pharmacokinetics of the HIV entry inhibitor CPT31 (cholesterol-PIE12-2-trimer) in healthy adults. This is a randomized, placebo-controlled, double-blind, single ascending dose study.

DETAILED DESCRIPTION:
This is a single subcutaneous (SC) dose study. Doses will be administered in an escalating manner following satisfactory review by a Protocol Safety Review Team (PSRT) of the safety, tolerability and pharmacokinetic (PK) data through Day 6 from the lower dose levels. 32 healthy subjects will be studied in 4 groups (Groups A1 to A4).

This study will comprise a placebo-controlled, double-blind, single-dose, sequential-group design in healthy subjects. Each subject will participate in 1 treatment period and reside in the Clinical Research Unit (CRU) from Day -1 through Day 6. It is planned for 6 subjects per dose level group to receive SC CPT31 and 2 subjects to receive matching placebo. Each group will be divided into 2 cohorts, with each cohort being dosed 72 hours apart. Sentinel dosing will take place in the first cohort, which will comprise 2 subjects, with 1 subject receiving CPT31 and 1 subject receiving placebo. The second cohort will comprise 6 subjects, with 5 subjects receiving CPT31 and 1 subject receiving placebo. Blood samples for PK analysis and assessment of immunogenicity will be collected predose and up to 5 days postdose, with an additional immunogenicity sample taken at the Follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, of any race, between 18 and 55 years of age, inclusive.
* Body mass index between 18.0 and 32.0 kg/m2, inclusive.
* In good health, determined by no clinically significant findings from medical and surgical history, physical examination, 12 lead ECG, vital signs measurements, and clinical laboratory evaluations (congenital nonhemolytic hyperbilirubinemia [e.g., suspicion of Gilbert's syndrome based on total and direct bilirubin] is not acceptable) at Screening and/or Day -1 as assessed by the Investigator (or designee).
* Females will not be pregnant or have been within the previous 3 months, or lactating, and females of childbearing potential and males will agree to use contraception.
* Able to comprehend and willing to sign an Informed Consent Form (ICF) and to abide by the study restrictions.

Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the Investigator (or designee).
* A ≥Grade 2 laboratory abnormality at Screening or Day -1 as defined by the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 dated July 2017.
* Estimated glomerular filtration rate (eGFR per CKD-Epi equation) of <90 ml/min/1.73 m2.
* Known sensitivity to CPT31 or any of its components.
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee).
* History of alcoholism or drug/chemical abuse within 2 years prior to Day -1.
* Alcohol consumption of > 21 units per week for males and > 14 units for females. One unit of alcohol equals 12 oz (360 mL) beer, 1½ oz (45 mL) liquor, or 5 oz (150 mL) wine.
* Positive urine drug screen at Screening or positive alcohol breath test result or positive urine drug screen on Day -1.
* Positive HIV test as documented by Combo Ag/Ab HIV 1/HIV-2 immunoassay.
* Positive hepatitis B surface antigen, positive hepatitis B core antibody with negative hepatitis B surface antibody test result, or positive hepatitis C antibody at Screening or within 3 months before first dose of study treatment.
* Participation in a clinical study involving administration of an investigational drug in the past 30 days prior to dosing.
* Use or intend to use any prescription or over the counter medications/products (including HIV medications being used for pre-exposure prophylaxis) other than hormone replacement therapy, oral, implantable, transdermal, injectable, or intrauterine contraceptives or acetaminophen up to 2 grams per day for no more than 3 consecutive days within 14 days prior to dosing, unless deemed acceptable by the Investigator (or designee).
* Use of tobacco or nicotine containing products within 3 months prior to Day -1, or positive cotinine at Screening or Day -1.
* Receipt of blood products within 2 months prior to Day -1.
* Donation of blood from 3 months prior to Screening, plasma from 2 weeks prior to Screening, or platelets from 6 weeks prior to Screening.
* Poor peripheral venous access.
* Have previously completed or withdrawn from this study or any other study investigating CPT31 and have previously received the investigational product.
* Subjects who, in the opinion of the Investigator (or designee), should not participate in this study.
* Have any clinically significant abnormal ECG results constituting a risk while taking the investigational product, as determined by the Investigator, such as any of the following, as determined by single 12-lead ECG: QT interval corrected for heart rate using Fridericia's method (QTcF) >450 ms for males and >470 ms for females, confirmed by calculating the mean of the original value and 2 repeats; QRS duration >120 ms confirmed by calculating the mean of the original value and 2 repeats; PR interval >220 ms confirmed by calculating the mean of the original value and 2 repeats; findings which would make QTc measurements difficult or QTc data uninterpretable; history of additional risk factors for torsades de pointes (e.g., heart failure, hypokalemia, family history of long QT syndrome); risks related to bradycardia, for example, second or third degree atrioventricular block or sick sinus syndrome.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2021-04-26 (Actual); Study Completion 2021-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan L Mueller, PhD, Study Director — Navigen, Inc.; Hugh A Coleman, DO, Principal Investigator — Covance
Locations (1):
- Covance Clinical Research Unit Inc., Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at a single site in the United States between 16 November 2020 (date of first informed consent) and 29 April 2021 (date of last subject's last assessment).
Pre-assignment Details: 32 subjects met inclusion criteria and were randomized to treatment.
Groups:
- Cohort 1 0.01 mg/kg CPT31: 6 subjects receiving a single subcutaneous injection of CPT31 (0.01 mg/kg)
  CPT31: CPT31 (cholesterol-PIE12-2-trimer) is a novel D-peptide HIV entry inhibitor that binds with high affinity to a conserved hydrophobic pocket within the gp41 trimer
- Cohort 2 0.04 mg/kg CPT31: 6 subjects receiving a single subcutaneous injection of CPT31 (0.04 mg/kg)
  CPT31: CPT31 (cholesterol-PIE12-2-trimer) is a novel D-peptide HIV entry inhibitor that binds with high affinity to a conserved hydrophobic pocket within the gp41 trimer
- Cohort 3 0.12 mg/kg CPT31: 6 subjects receiving a single subcutaneous injection of CPT31 (0.12 mg/kg) CPT31: CPT31 (cholesterol-PIE12-2-trimer) is a novel D-peptide HIV entry inhibitor that binds with high affinity to a conserved hydrophobic pocket within the gp41 trimer
- Cohort 4 0.24 mg/kg CPT31: 6 subjects receiving a single subcutaneous injection of CPT31 (0.24 mg/kg)
  CPT31: CPT31 (cholesterol-PIE12-2-trimer) is a novel D-peptide HIV entry inhibitor that binds with high affinity to a conserved hydrophobic pocket within the gp41 trimer
- Placebo: 8 subjects receiving a single subcutaneous placebo injection
Period: Overall Study
Arm/Group | Cohort 1 0.01 mg/kg CPT31 | Cohort 2 0.04 mg/kg CPT31 | Cohort 3 0.12 mg/kg CPT31 | Cohort 4 0.24 mg/kg CPT31 | Placebo
Started | 6 | 6 | 6 | 6 | 8
Completed | 5 | 6 | 6 | 6 | 8
Not Completed | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1 0.10 mg/kg CPT31: 6 subjects receiving a single subcutaneous injection of CPT31 (0.01 mg/kg)
  CPT31: CPT31 (cholesterol-PIE12-2-trimer) is a novel D-peptide HIV entry inhibitor that binds with high affinity to a conserved hydrophobic pocket within the gp41 trimer
- Total: Total of all reporting groups
Arm/Group | Cohort 1 0.10 mg/kg CPT31 | Cohort 2 0.04 mg/kg CPT31 | Cohort 3 0.12 mg/kg CPT31 | Cohort 4 0.24 mg/kg CPT31 | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 6 | 6 | 8 | 32
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.0 (11.26) | 41.8 (9.28) | 25.2 (10.25) | 38.7 (11.08) | 38.5 (10.77) | 37.1 (11.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 2 | 1 | 2 | 11
  Male | 3 | 3 | 4 | 5 | 6 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4 | 3 | 5 | 16
  Not Hispanic or Latino | 5 | 3 | 2 | 3 | 3 | 16
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 4 | 2 | 1 | 2 | 12
  White | 3 | 1 | 4 | 5 | 6 | 19
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 6 | 6 | 8 | 32
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — body mass index (kg/m2)
  kg/m^2 | 24.32 (5.426) | 27.08 (2.567) | 23.45 (3.026) | 25.47 (2.233) | 25.00 (2.898) | 25.06 (3.380)

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: Number of subjects experiencing serious adverse events (SAEs)
Time Frame: Check-in (Day -1) through Follow-up (Day 28-30)
Population: The safety population included all subjects who received at least 1 dose of study treatment (CPT31 or placebo).
Measure: Number; unit: participants experiencing adverse events
Arm/Group | Cohort 1 0.01 mg/kg CPT31 | Cohort 2 0.04 mg/kg CPT31 | Cohort 3 0.12 mg/kg CPT31 | Cohort 4 0.24 mg/kg CPT31 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
participants experiencing adverse events | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Cmax
Description: maximum observed plasma concentration (ng/mL)
Time Frame: Day 1 predose, 0.5 h, 1 h, 2 h, 4 h, 6 h, 8 h, 10 h, 12 h, 16 h, Day 2 (24 h), Day 3 (48 h), Day 4 (72 h), Day 5 (96 h), and Day 6 (120 h)
Population: The pharmacokinetic (PK) population included all subjects who received at least 1 dose of CPT31 and had evaluable PK data.
Measure: Mean (Full Range); unit: ng/mL
Arm/Group | Cohort 1 0.01 mg/kg CPT31 | Cohort 2 0.04 mg/kg CPT31 | Cohort 3 0.12 mg/kg CPT31 | Cohort 4 0.24 mg/kg CPT31
Number analyzed (Participants) | 5 | 6 | 6 | 6
ng/mL | 27.6 [22.7 to 39.4] | 91.0 [45.1 to 144] | 247 [147 to 487] | 666 [393 to 1930]
Statistical Analysis 1: Comparison: Cohort 1 0.01 mg/kg CPT31 vs Cohort 2 0.04 mg/kg CPT31 vs Cohort 3 0.12 mg/kg CPT31 vs Cohort 4 0.24 mg/kg CPT31; CPT31 dose proportionality will be examined across dose groups using a power model approach or ANOVA model, as appropriate.PK parameters will be analyzed using a power model that will have the following form: parameter = intercept × dose^slope + random error. Using the natural log (ln) transformation, a power model can be expressed as a linear regression equation: ln(parameter) = intercept + slope × ln(dose) + random error. For dose proportionality, the slope = 1; for dose independence, = 0; Test type: Other; p < 0.05, ANOVA

3. Secondary Outcome: Tmax
Description: time of maximum observed plasma concentration (h)
Time Frame: as for outcome 2
Population: The PK population included all subjects who received at least 1 dose of CPT31 and had evaluable PK data.
Measure: Median (Full Range); unit: Hours post administration
Groups:
- Cohort 4 0.24 mg/kg CPT3: 6 subjects receiving a single subcutaneous injection of CPT31 (0.24 mg/kg)
  CPT31: CPT31 (cholesterol-PIE12-2-trimer) is a novel D-peptide HIV entry inhibitor that binds with high affinity to a conserved hydrophobic pocket within the gp41 trimer
Arm/Group | Cohort 1 0.01 mg/kg CPT31 | Cohort 2 0.04 mg/kg CPT31 | Cohort 3 0.12 mg/kg CPT31 | Cohort 4 0.24 mg/kg CPT3
Number analyzed (Participants) | 5 | 6 | 6 | 6
Hours post administration | 6.00 [4.00 to 12.0] | 7.00 [4.00 to 16.0] | 7.00 [4.00 to 10.00] | 4.00 [0.500 to 24.00]
Statistical Analysis 1: Comparison: Cohort 1 0.01 mg/kg CPT31 vs Cohort 2 0.04 mg/kg CPT31 vs Cohort 3 0.12 mg/kg CPT31 vs Cohort 4 0.24 mg/kg CPT3; [analysis description as in outcome 2, analysis 1]; Test type: Other; p < 0.05, ANOVA

4. Secondary Outcome: T1/2
Description: apparent plasma terminal elimination half-life (h)
Time Frame: as for outcome 2
Population: Insufficient data for Cohorts 1&2. No t1/2 estimate possible for 3 subjects in Cohorts 1&2, and 1 in Cohort 4 as a reliable regression could not be fitted to the data. Per SAP: terminal elimination rate constant (λz) will only be calculated when a reliable estimate is obtained using ≥3 data points, and adjusted coefficient for determination of exponential fit (R2-adj) of the regression line is ≥0.7. Parameters requiring λz will only be calculated if R2-adj value of the regression is ≥0.7.
Measure: Mean (Full Range); unit: Hours post administration
Arm/Group | Cohort 1 0.01 mg/kg CPT31 | Cohort 2 0.04 mg/kg CPT31 | Cohort 3 0.12 mg/kg CPT31 | Cohort 4 0.24 mg/kg CPT31
Number analyzed (Participants) | 5 | 6 | 6 | 5
Hours post administration | NA [NA to NA] — One subject in Cohort 1 displayed plasma concentrations below the limit of quantification at all timepoints. No t1/2 estimate was possible for 3 subjects in Cohort 1, 3 subjects in Cohort 2, and 1 subject in cohort 4 because a reliable regression could not be fitted to the data. | NA [NA to NA] — One subject in Cohort 1 displayed plasma concentrations below the limit of quantification at all timepoints. No t1/2 estimate was possible for 3 subjects in Cohort 1, 3 subjects in Cohort 2, and 1 subject in cohort 4 because a reliable regression could not be fitted to the data. | 17.2 [14.2 to 20.8] | 15.2 [12.7 to 19.2]
Statistical Analysis 1: Comparison: Cohort 1 0.01 mg/kg CPT31 vs Cohort 2 0.04 mg/kg CPT31 vs Cohort 3 0.12 mg/kg CPT31 vs Cohort 4 0.24 mg/kg CPT31; The lack of fit test will be conducted for the statistical assessment of linearity assumption (AOL), and thus appropriateness of a power model. PK parameter is dose proportional if AOL is ruled acceptable and the 95% confidence interval for the slope spans 1. If the AOL is ruled unacceptable for any PK parameter, its corresponding PK parameter normalized by dose administered will be ln-transformed and analyzed using an analysis of variance (ANOVA) model. The model will include dose as a factor; Test type: Other; p < 0.05, Regression, Linear

5. Secondary Outcome: Area Under the Concentration Curve (AUC) 0-∞
Description: area under the concentration versus time curve (AUC) from time zero to infinity (h*ng/mL)
Time Frame: as for outcome 2
Population: Insufficient data for Cohorts 1&2. No (AUC)0-∞ estimate possible for 3 subjects in Cohorts 1&2, and 1 in Cohort 4 as a reliable regression could not be fitted to the data. Per SAP: terminal elimination rate constant (λz) will only be calculated when a reliable estimate is obtained using ≥3 data points, and adjusted coefficient for determination of exponential fit (R2-adj) of the regression line is ≥0.7. Parameters requiring λz will only be calculated if R2-adj value of the regression is ≥0.7.
Measure: Mean (Full Range); unit: h*ng/mL
Arm/Group | Cohort 1 0.01 mg/kg CPT31 | Cohort 2 0.04 mg/kg CPT31 | Cohort 3 0.12 mg/kg CPT31 | Cohort 4 0.24 mg/kg CPT31
Number analyzed (Participants) | 5 | 6 | 6 | 6
h*ng/mL | NA [NA to NA] — One subject in Cohort 1 displayed plasma concentrations below the limit of quantification at all timepoints. No t1/2 estimate was possible for 3 subjects in Cohort 1, 3 subjects in Cohort 2, and 1 subject in cohort 4 because a reliable regression could not be fitted to the data. | NA [NA to NA] — One subject in Cohort 1 displayed plasma concentrations below the limit of quantification at all timepoints. No t1/2 estimate was possible for 3 subjects in Cohort 1, 3 subjects in Cohort 2, and 1 subject in cohort 4 because a reliable regression could not be fitted to the data. | 8170 [6300 to 10900] | 21200 [15400 to 28100]
Statistical Analysis 1: Comparison: Cohort 1 0.01 mg/kg CPT31 vs Cohort 2 0.04 mg/kg CPT31 vs Cohort 3 0.12 mg/kg CPT31 vs Cohort 4 0.24 mg/kg CPT31; The lack of fit test will be conducted for the statistical assessment of linearity assumption (AOL), and thus appropriateness of a power model. PK parameter is dose proportional if AOL is ruled acceptable and the 95% CI for the slope spans 1. If the AOL is ruled unacceptable for any PK parameter, its corresponding PK parameter normalized by dose administered will be ln-transformed and analyzed using an analysis of variance (ANOVA) model. The model will include dose as a factor; Test type: Other; p < 0.05, Regression, Linear

6. Secondary Outcome: AUC0-tlast
Description: area under the concentration versus time curve (AUC) from time zero to time of the last quantifiable concentration (h*ng/mL)
Time Frame: as for outcome 2
Population: The PK population included all subjects who received at least 1 dose of CPT31 and had evaluable PK data.
Measure: Mean (Full Range); unit: h*ng/mL
Arm/Group | Cohort 1 0.01 mg/kg CPT31 | Cohort 2 0.04 mg/kg CPT31 | Cohort 3 0.12 mg/kg CPT31 | Cohort 4 0.24 mg/kg CPT31
Number analyzed (Participants) | 5 | 6 | 6 | 6
h*ng/mL | 253 [156 to 453] | 1660 [919 to 2420] | 7000 [4870 to 10500] | 19500 [14500 to 27200]
Statistical Analysis 1: Comparison: Cohort 1 0.01 mg/kg CPT31 vs Cohort 2 0.04 mg/kg CPT31 vs Cohort 3 0.12 mg/kg CPT31 vs Cohort 4 0.24 mg/kg CPT31; [analysis description as in outcome 5, analysis 1]; Test type: Other; p < 0.05, Regression, Linear

7. Secondary Outcome: Total Plasma Clearance (CL/F)
Description: apparent total plasma clearance (L/h/kg)
Time Frame: as for outcome 2
Population: Insufficient data for Cohorts 1&2. No CL/F estimate possible for 3 subjects in Cohorts 1&2, and 1 in Cohort 4 as a reliable regression could not be fitted to the data. Per SAP: terminal elimination rate constant (λz) will only be calculated when a reliable estimate is obtained using ≥3 data points, and adjusted coefficient for determination of exponential fit (R2-adj) of the regression line is ≥0.7. Parameters requiring λz will only be calculated if R2-adj value of the regression is ≥0.7
Measure: Mean (Full Range); unit: L/h/kg
Arm/Group | Cohort 1 0.01 mg/kg CPT31 | Cohort 2 0.04 mg/kg CPT31 | Cohort 3 0.12 mg/kg CPT31 | Cohort 4 0.24 mg/kg CPT31
Number analyzed (Participants) | 5 | 6 | 6 | 6
L/h/kg | NA [NA to NA] — One subject in Cohort 1 displayed plasma concentrations below the limit of quantification at all timepoints. No t1/2 estimate was possible for 3 subjects in Cohort 1, 3 subjects in Cohort 2, and 1 subject in cohort 4 because a reliable regression could not be fitted to the data. | NA [NA to NA] — One subject in Cohort 1 displayed plasma concentrations below the limit of quantification at all timepoints. No t1/2 estimate was possible for 3 subjects in Cohort 1, 3 subjects in Cohort 2, and 1 subject in cohort 4 because a reliable regression could not be fitted to the data. | 17.2 [14.2 to 20.8] | 15.2 [12.7 to 19.2]
Statistical Analysis 1: Comparison: Cohort 1 0.01 mg/kg CPT31 vs Cohort 2 0.04 mg/kg CPT31 vs Cohort 3 0.12 mg/kg CPT31 vs Cohort 4 0.24 mg/kg CPT31; [analysis description as in outcome 5, analysis 1]; Test type: Other; p < 0.05, Regression, Linear

8. Secondary Outcome: Vz/F
Description: apparent volume of distribution (L/kg)
Time Frame: as for outcome 2
Population: Insufficient data for Cohorts 1&2. No Vz/F estimate possible for 3 subjects in Cohorts 1&2, and 1 in Cohort 4 as a reliable regression could not be fitted to the data. Per SAP: terminal elimination rate constant (λz) will only be calculated when a reliable estimate is obtained using ≥3 data points, and adjusted coefficient for determination of exponential fit (R2-adj) of the regression line is ≥0.7. Parameters requiring λz will only be calculated if R2-adj value of the regression is ≥0.7
Measure: Mean (Full Range); unit: L/kg
Arm/Group | Cohort 1 0.01 mg/kg CPT31 | Cohort 2 0.04 mg/kg CPT31 | Cohort 3 0.12 mg/kg CPT31 | Cohort 4 0.24 mg/kg CPT31
Number analyzed (Participants) | 5 | 6 | 6 | 6
L/kg | NA [NA to NA] — Insufficient data for Cohorts 1 and 2 | NA [NA to NA] — Insufficient data for Cohorts 1 and 2 | 0.365 [0.240 to 0.571] | 0.248 [0.192 to 0.431]
Statistical Analysis 1: Comparison: Cohort 1 0.01 mg/kg CPT31 vs Cohort 2 0.04 mg/kg CPT31 vs Cohort 3 0.12 mg/kg CPT31 vs Cohort 4 0.24 mg/kg CPT31; [analysis description as in outcome 5, analysis 1]; Test type: Other; p < 0.05, Regression, Linear

9. Secondary Outcome: Ae
Description: amount of drug excreted in the urine (ng/mL)
Time Frame: as for outcome 2
Population: Concentrations for all subjects in Cohorts 1-3 were below the limit of quantitation. Urine was not collected for Cohort 4.
Measure: Mean (Full Range); unit: ng/mL
Arm/Group | Cohort 1 0.01 mg/kg CPT31 | Cohort 2 0.04 mg/kg CPT31 | Cohort 3 0.12 mg/kg CPT31 | Cohort 4 0.24 mg/kg CPT31
Number analyzed (Participants) | 5 | 6 | 6 | 0
ng/mL | NA [NA to NA] — Concentrations for all subjects in Cohorts 1-3 were below the limit of quantitation. | NA [NA to NA] — Concentrations for all subjects in Cohorts 1-3 were below the limit of quantitation. | NA [NA to NA] — Concentrations for all subjects in Cohorts 1-3 were below the limit of quantitation. |
Statistical Analysis 1: Comparison: Cohort 1 0.01 mg/kg CPT31 vs Cohort 2 0.04 mg/kg CPT31 vs Cohort 3 0.12 mg/kg CPT31; Concentrations for all subjects in Cohorts 1-3 were below the limit of quantification; Test type: Other; p < 0.05, Regression, Linear

10. Secondary Outcome: Fe
Description: percentage of dose excreted unchanged in the urine (%)
Time Frame: as for outcome 2
Population: as for outcome 9
Measure: Mean (Full Range); unit: percentage of drug excreted unchanged
Arm/Group | Cohort 1 0.01 mg/kg CPT31 | Cohort 2 0.04 mg/kg CPT31 | Cohort 3 0.12 mg/kg CPT31 | Cohort 4 0.24 mg/kg CPT31
Number analyzed (Participants) | 5 | 6 | 6 | 0
percentage of drug excreted unchanged | NA [NA to NA] — Concentrations for all subjects in Cohorts 1-3 were below the limit of quantitation. | NA [NA to NA] — Concentrations for all subjects in Cohorts 1-3 were below the limit of quantitation. | NA [NA to NA] — Concentrations for all subjects in Cohorts 1-3 were below the limit of quantitation. |
Statistical Analysis 1: Comparison: Cohort 1 0.01 mg/kg CPT31 vs Cohort 2 0.04 mg/kg CPT31 vs Cohort 3 0.12 mg/kg CPT31; Concentrations for all subjects in Cohorts 1-3 were below the limit of quantitation; Test type: Other; p < 0.05, Regression, Linear

11. Secondary Outcome: Renal Clearance (CLR)
Description: renal clearance (L/h/kg)
Time Frame: as for outcome 2
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: L/h/kg
Arm/Group | Cohort 1 0.01 mg/kg CPT31 | Cohort 2 0.04 mg/kg CPT31 | Cohort 3 0.12 mg/kg CPT31 | Cohort 4 0.24 mg/kg CPT31
Number analyzed (Participants) | 5 | 6 | 6 | 0
L/h/kg | NA (NA) — Concentrations for all subjects in Cohorts 1-3 were below the limit of quantitation. | NA (NA) — Concentrations for all subjects in Cohorts 1-3 were below the limit of quantitation. | NA (NA) — Concentrations for all subjects in Cohorts 1-3 were below the limit of quantitation. |
Statistical Analysis 1: Comparison: Cohort 1 0.01 mg/kg CPT31 vs Cohort 2 0.04 mg/kg CPT31 vs Cohort 3 0.12 mg/kg CPT31; Concentrations for all subjects in Cohorts 1-3 were below the limit of quantitation; Test type: Other; p < 0.05, Regression, Linear

12. Secondary Outcome: Immunogenicity
Description: Number of subjects with measurable levels of anti-CPT31 antibodies in serum
Time Frame: Pre-dose on Day 1 through Follow-up (Day 28-30)
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 0.01 mg/kg CPT31 | Cohort 2 0.04 mg/kg CPT31 | Cohort 3 0.12 mg/kg CPT31 | Cohort 4 0.24 mg/kg CPT31 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
Participants | 0 | 0 | 1 | 0 | 0
Statistical Analysis 1: Comparison: Cohort 1 0.01 mg/kg CPT31 vs Cohort 2 0.04 mg/kg CPT31 vs Cohort 3 0.12 mg/kg CPT31 vs Cohort 4 0.24 mg/kg CPT31; [analysis description as in outcome 5, analysis 1]; Test type: Other; p < 0.05, Regression, Linear

ADVERSE EVENTS:
Time Frame: 30 days
Description: Subjects will be observed for any signs or symptoms and asked about their condition by open questioning. Subjects will also be encouraged to spontaneously report adverse events (AEs) occurring at any other time during the study. All nonserious AEs, whether reported by the subject voluntarily or upon questioning, or noted on physical examination, will be recorded from initiation of study drug until study end. Serious AEs will be recorded from signing the informed consent form until study end.
Arm/Group | Cohort 1 0.01 mg/kg CPT31 | Cohort 2 0.04 mg/kg CPT31 | Cohort 3 0.12 mg/kg CPT31 | Cohort 4 0.24 mg/kg CPT31 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/8
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 2/6 | 5/6 | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 0.01 mg/kg CPT31 (N=6) | Cohort 2 0.04 mg/kg CPT31 (N=6) | Cohort 3 0.12 mg/kg CPT31 (N=6) | Cohort 4 0.24 mg/kg CPT31 (N=6) | Placebo (N=8)
Injection Site Erythema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 0 (0)
Injection Site Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Injection Site Induration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Injection Site Pruritis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-07-27): https://cdn.clinicaltrials.gov/large-docs/83/NCT04672083/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-13): https://cdn.clinicaltrials.gov/large-docs/83/NCT04672083/SAP_001.pdf